CLINICAL TRIAL: NCT00362037
Title: Irbesartan In Hypertensive Patients With Left Ventricular Hypertrophy
Brief Title: I SELECT - Irbesartan In Hypertensive Patients With Left Ventricular Hypertrophy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM_L_0255
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Irbesartan (Aprovel) — Aprovel (150 & 300mg) & CoAprovel (300/12.5mg hydrochlorothiazide one per day per os.

SUMMARY:
* To evaluate Blood Pressure (BP) reduction to the targeted values (BP ≤ 140/90 mm Hg in non-diabetic patients, and ≤ 130/80 mm Hg in diabetic patients).
* To emphasize and to evaluate the benefit of Irbesartan in the reduction of left ventricular mass index in hypertensive patients with left ventricular hypertrophy.
* To demonstrate safety of Irbesartan in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven mild to moderate Hypertension.
* Patients must have left ventricular mass index > 130g/m2 in men, > 100g/m2 in women, as evidenced by echocardiography before inclusion.
* Newly diagnosed "naïve" hypertensive patients (no prior treatment for hypertension). OR,
* Patients who were receiving antihypertensive agents (maximum two agents including one diuretic) with blood pressure targets achieved, yet, in the investigator's opinion, those patients would benefit more from switching to the study medication. These patients will undergo a wash out period for not less than 7 days prior to enrollment.

Exclusion Criteria:

* Severe hypertension (Systolic BP ≥ 180 mm Hg or Diastolic BP ≥ 110 mm Hg).
* Patients with left ventricular ejection fraction < 45%.
* Patients with severe left ventricular hypertrophy.
* Patients with known secondary hypertension (for another cause other than type 2 Diabetes Mellitus).
* Diabetic patients with HbA1c > 10%.
* Significant chronic renal impairment (Serum creatinine > 2.0 mg/dL).
* Significant liver disease as shown by SGPT/SGOT (ALT/AST) > 2.5 times the upper limit of the normal range.
* Currently pregnant or lactating females.
* Women of childbearing potential not protected by effective contraceptive method of birth control and/or who are unwilling or unable to be tested for pregnancy.
* Any patient who is in need for a combination antihypertensive therapy from the start (from the medical point of view of his/her physician).
* Known hypersensitivity to irbesartan, other ARBs(Angiotensin Receptor Blockers), hydrochlorothiazide, or other thiazide diuretics.
* Patients with malignancy during the past 5 years, known collagen disease or severe cardiac, cerebrovascular or gastric disease.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2006-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Reduction in BP to target values according to the ESC 2003 Hypertension Guidelines | During the study conduct
Reduction in left ventricular hypertrophy from baseline values to week 36. | during the study conduct

SECONDARY OUTCOMES:
Occurrence of any side effect leading to treatment discontinuation. | During all the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Mosaad I Morsi, MBBCh, MSc, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Cairo, Egypt